CLINICAL TRIAL: NCT04340206
Title: The Effectiveness of the Youth Compass Plus: The Novel Five-week Web- and Mobile-based Acceptance- and Commitment Therapy Program to Promote Adolescent Psychological Flexibility and Well-being
Brief Title: Youth Compass Plus
Acronym: YouthCompass+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jyvaskyla (Other)
Collaborators: Academy of Finland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 324638
Record Dates: First submitted 2020-04-01; First posted 2020-04-09 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Psychological Flexibility; Psychological Well-being
Keywords: Adolescents; Acceptance Commitment Therapy; Web- and mobile-based intervention; Psychological flexibility; Psychological well-being; Career preparation; Successful educational transitions
MeSH Terms: conditions — Psychological Well-Being | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Efficacy study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- face-to-face support and Chatbot online support group (Experimental): Experimental, Intervention Group A: face-to-face support and Chatbot online support group: 5-week intervention according to ACT principles with the web- and mobile-based Youth Compass plus program, face-to-face support (2 meetings) and weekly online support and feedback from the Chabot eCoach built within the program (one third of the participants is randomly assigned to this group)
  Interventions: Behavioral: face-to-face support and Chatbot online support group
- only chat-robot online support group (Experimental): Experimental, Intervention Group B: only chat-robot online support group: 5-week intervention according to ACT principles with the web-and mobile-based Youth Compass plus program, no face-to-face support, and weekly online support and feedback from the chatbot eCoach built within the program (one third of the participants is randomly assigned to this group)
  Interventions: Behavioral: only chat-robot online support group
- Experimental Control (Experimental): Experimental Control:
  Control group, no intervention (one third of the participants is randomly assigned to this group)
  Interventions: Behavioral: Control group, no intervention

INTERVENTIONS:
Behavioral: face-to-face support and Chatbot online support group — Behavioral: Structured web- and mobile-based intervention with Youth Compass plus program to support adolescents' psychological flexibility, well-being, and subsequently support successful transition to upper secondary education. The Youth Compass plus is a five-week online program aiming to enhance adolescents' psychological flexibility by guiding adolescents in exploring their values and setting goals and changing behaviors according to their goals (week 1), and learning acceptance, defusion and mindfulness skills (weeks 2-3) and integrating these skills into their personal and social life (weeks 4-5). The participants in this condition receive weekly online support and feedback from the eCoach built within the program. In addition, they meet and get support from their human coach (i.e., psychology student) twice in the face-to-face meetings.
  Arms: face-to-face support and Chatbot online support group
Behavioral: only chat-robot online support group — Behavioral: Structured web- and mobile-based intervention with Youth Compass plus program to adolescents' psychological flexibility, well-being, and subsequently support successful transition to upper secondary education. The Youth Compass plus is a five-week online program aiming to enhance adolescents' psychological flexibility by guiding adolescents in exploring their values and setting goals and changing behaviors according to their goals (week 1), and learning acceptance, defusion and mindfulness skills (weeks 2-3) and integrating these skills into their personal and social life (weeks 4-5). The participants in this condition receive weekly online support and feedback from the eCoach built within the program.
  Arms: only chat-robot online support group
Behavioral: Control group, no intervention — Behavioral: No intervention
  Arms: Experimental Control

SUMMARY:
The aim of this randomized control trial is to examine the effectiveness of a novel web- and mobile-based Acceptance and Commitment Therapy program (Youth Compass plus) to promote adolescents' psychological flexibility and well-being and subsequently support their successful transition from basic education to upper secondary education. Our aim is also to compare the efficacy of Youth Compass plus using either an eCoach providing automated personal support to the user or an eCoach and a Human Coach providing personal support to the user. Additionally, we will investigate whether the efficacy of the Youth Compass plus varies according to different individual and contextual factors.

Using the internet to deliver interventions is assumed to be particularly motivating for youth who enjoy spending time online using different social media. Web-based interventions have several advantages; they can include more information and treatment components than traditionally delivered treatments and they are accessible at any time and place. The five-week structured intervention is delivered using the novel web- and mobile-based program Youth Compass plus. Youth Compass plus has been developed based on the feedback for the Youth COMPASS pilot program (see ClinicalTrials.gov, NCT03274934). The exercises of Youth Compass plus have been modified, visual aspects have been improved and new game-based interactive elements have been developed. In the Youth COMPASS pilot study, psychology students acted as (human) coaches for the users. While interaction with a personal coach increases commitment to the program, the need to train and supervise coaches limits large scale dissemination. To provide an alternative that is less demanding in terms of resources, we have developed a chatbot (eCoach) as a new feature within the new Youth Compass plus program. The automated eCoach provides personal support within the program and via text messages. The eCoach provides support and encouragement, reminds about using Youth Compass plus, sends individualized feedback, and recommends different exercises.

DETAILED DESCRIPTION:
The aim of this randomized trial is to examine whether Youth Compass plus enhances adolescents' (a) psychological skills, particularly with respect to finding a purpose, and psychological flexibility and adaptation skills as the ACT process outcomes; (b) career preparation and psychological well-being as the proximal outcomes; and (c) the initiation of upper secondary education studies and engagement in upper secondary education as the distal outcomes.

In addition, our aim is to investigate the ACT processes and mediating mechanisms of the Youth Compass plus program, and to explore the extent to which the effectiveness of the Youth Compass plus varies according to the differences in various individual and contextual factors.

H1: The study expects that the Youth Compass plus is more effective than no intervention. Youth Compass plus is expected to promote ACT proximal youth outcomes, as well as the youth distal outcomes.

H2: In addition, the study expects that the Youth Compass plus will promote the distal outcomes through enhancing the ACT process outcomes and the proximal outcomes.

H3: The study expects that Youth Compass plus is more effective for those adolescents who accept the intervention well, take part intensively and diversely in different exercises, as well as among the adolescents who are initially highly emotionally reactive.

ELIGIBILITY:
Inclusion and Exclusion Criteria:

Approximately 600-1000 Finnish 14-16 year old adolescents from non-clinical school-age population will fill in a pre-questionnaire. Based on this data the participants for the randomized control trial will be selected from the two gender-balanced groups of Finnish adolescents:

1. Adolescents (n = 150) who have heightened (pre-clinical) level of symptoms of stress/anxiety/depression in the screening measures (no diagnosis is required for participation).
2. Randomly chosen adolescents (n=150) who have no symptoms of stress/anxiety/depression in the screening measures

Adolescents from both groups are randomly assigned in three conditions: (a) five weeks of Youth Compass plus with support from chatbot + face-to-face support (altogether two face-to-face meetings); b) five-weeks of Youth Compass plus with support from chatbot only; or (c) no intervention. At the baseline (fall 2020) the participants will be ninth-graders facing the transition to upper secondary education.

Ages: 14 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 348 (Actual)
Dates: Start 2020-09-08 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
psychological flexibility | Change from baseline at 2 and 6 months after the intervention
  Comprehensive assessment of Acceptance and Commitment Therapy processes, CompACT; Francis et al., 2016
psychological flexibility | Change from baseline at 2 and 6 months after the intervention
  Cognitive Fusion Questionnaire (Gillanders et al., 2014)
life satisfaction | Change from baseline at 2 and 6 months after the intervention
  Satisfaction with Life Scale, SWLS, Diener et al., 1985
mental well-being | Change from baseline at 2 and 6 months after the intervention
  Warwick-Edinburgh Mental Well-being Scale WEMWBS; THL 2011
stress symptoms | Change from baseline at 2 and 6 months after the intervention
  Perceived Stress Scale, PSS-10; Cohen et al., 1983
anxiety symptoms | Change from baseline at 2 and 6 months after the intervention
  short-form of the state scale of the Spielberger State-Trait Anxiety Inventory, STAI; Marteau & Becker, 1992
depressive symptoms | Change from baseline at 2 and 6 months after the intervention
  Depression Scale, DEPS; Salokangas et al., 1995
Career choice preparedness | Change from baseline at 2 and 6 months after the intervention
  career choice self-efficacy, career-related insecurity, preparation against setbacks, Koivisto et al., 2011

SECONDARY OUTCOMES:
perfectionism | Change from baseline at 2 and 6 months after the intervention
  The Child-Adolescent; Perfectionism Scale, CAPS; Gordon et al., 2016
self-compassion | Change from baseline at 2 and 6 months after the intervention
  Self-Compassion Scale - Short Form; Raes et al., 2011
prosocial aspirations | Change from baseline at 2 and 6 months after the intervention
  short form of the Aspirations Index, Marshall, 2019
academic buoyancy | Change from baseline at 2 and 6 months after the intervention
  short Academic buoyancy scale; Martin & Marsh, 2008
school well-being | Change from baseline at 2 and 6 months after the intervention
  school satisfaction, anti-school attitude, school-related stress, WHO
academic performance | Change from baseline at 2 and 6 months after the intervention
  grade point average
truancy and school absences | Change from baseline at 2 and 6 months after the intervention
  truancy and school absences, Finnish School Health Questionnaire
educational attainment, information from school registers | 2020-2025 (not possible to provide more specitic time frame)
  initiation of upper secondary education, progress in studies, changes in study field, graduation time,

OTHER OUTCOMES:
learning-related expectations and behaviours | Change from baseline at 2 and 6 months after the intervention
  success expectations, task-focused behavior and planning; Nurmi et al., 1995
educational expectations | Change from baseline at 2 and 6 months after the intervention
  educational expectations
quality of close relationships | Change from baseline at 2 and 6 months after the intervention
  conflict and closeness in child-parent, child-teacher, and child-best relationships (Pianta)
personality | Change from baseline at 2 and 6 months after the intervention
  short Big Five, Gostling et al., 2003)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychology University of Jyvaskyla, Jyväskylä, Finland

IPD SHARING:
Plan to Share IPD: No
Ownership of the data will reside with the University of Jyväskylä and the data are managed by the PI and her research team. Research co-operation agreements will be made with the collaborators about confidentiality issues, data management principles, and use of data in publications. Other researchers are encouraged to use the data; however, it requires a research plan and the permission of the research team. Principally, the PI or someone else from the research team will be one of the co-authors in all publications written from the data.